CLINICAL TRIAL: NCT03540472
Title: Tacrolimus Treatment for Refractory Pure Red Cell Aplasia, a Prospective Study
Brief Title: Tacrolimus Treatment for Refractory PRCA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tacrolimus-001
Record Dates: First submitted 2018-05-14; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Pure Red Cell Aplasia
Keywords: tacrolimus; refractory pure red cell aplasia; prospective study
MeSH Terms: conditions — Red-Cell Aplasia, Pure | interventions — Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- efficiency of tacrolimus on PRCA (Experimental): A prospective research of the tacrolimus efficiency on refractory PRCA patients On refractory PRCA patients, tacrolimus was tried. Dosage: 1mg bid and tacrolimus trough targets were 5-10 ng/ml throughout the study.
  Medication time should last at least 6 months.
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — On refractory PRCA patients, tacrolimus was tried. Dosage: 1mg bid and tacrolimus trough targets were 5-10 ng/ml throughout the study
  Other Names: tacrolimus capsule

SUMMARY:
Pure red cell aplasia (PRCA) is a kind of anemia characterized by severe reticulocytopenia and obvious bone marrow erythroblastic cells decreased. Cyclosporine and /or steroids are the first line therapy but some patients were refractory or intolerance to the treatment. The effects of the second line therapy are also not satisfactory and sometimes not available. The investigators aim to explore the efficacy and side-effect of tacrolimus for refractory PRCA.

DETAILED DESCRIPTION:
Pure red cell aplasia (PRCA) is a rare normocytic normochromic anemia with reticulocytopenia, characterized by a reduction of erythroid precursors from the bone marrow, could be divided into congenital and acquired PRCA according to pathogenesis. Congenital PRCA, also known as Diamond-Blackfan syndrome, has been associated with pathogenic variant in GATA1 and TSR2 and gene encode ribosomal proteins. Acquired PRCA can be a primary disease which is usually mediated by immunology, or secondary to other diseases, such as lymphoproliferative diseases, autoimmune diseases, thymoma, infection, or drugs. The first line therapy of acquired PRCA is Cyclosporine A and steroids, the second line therapy are anti-CD20, ATG, immunosuppressive drugs like cyclophosphamide, bone marrow transplantation. Unfortunately, some patients did not response or tolerate the above treatments. Tacrolimus, also known as FK506, is an agent mainly used after allogeneic organ transplant to lower risk of organ rejection. Tacrolimus could inhibit the production the production of IL-2, and also used in the therapy of other T cell mediated diseases. Tacrolimus primarily has been approved for prevent organ transplant rejection, especially in renal transplantation, tacrolimus also promises to treat autoimmune, degenerative and hyperproliferative disorders. Recently, tacrolimus has been reported to be effective and well tolerated for many immune-mediated cytopenias, such as autoimmune lymphoproliferative syndrome, immune thrombocytopenia, EVANS syndrome, etc. However, due to the rare occurrence of PRCA and good response rate to cyclosporine, there are very few studies of tacrolimus on refractory PRCA so far. In this study, it is anticipate to evaluate the effect of tacrolimus on 30 patients with refractory PRCA, the side-effects was documented and plasma concentration of tacrolimus will be monitor.

ELIGIBILITY:
Inclusion Criteria:

Refractory pure red cell aplasia. 18-80 years old. No response or intolerant to first and second line therapies. Written informed consent.

Exclusion Criteria:

Other diseases which might cause hematological abnormalities. Response and well tolerate to first or second line therapy. Patients who are under 18-year-old or over 80-year-old. Pregnant or lactating. Patients unwilling to or unable to comply with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-10 (Estimated); Primary Completion 2018-12-10 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | 6 months
  Hemoglobin level in g/L

SECONDARY OUTCOMES:
Hemoglobin level | 2 years
  Hemoglobin level in g/L

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Langer RM, Hene R, Vitko S, Christiaans M, Tedesco-Silva H Jr, Ciechanowski K, Cassuto E, Rostaing L, Vilatoba M, Machein U, Ulbricht B, Junge G, Dong G, Pascual J. Everolimus plus early tacrolimus minimization: a phase III, randomized, open-label, multicentre trial in renal transplantation. Transpl Int. 2012 May;25(5):592-602. doi: 10.1111/j.1432-2277.2012.01465.x. Epub 2012 Mar 26. PMID 22471345
- [Result] Patsenker E, Schneider V, Ledermann M, Saegesser H, Dorn C, Hellerbrand C, Stickel F. Potent antifibrotic activity of mTOR inhibitors sirolimus and everolimus but not of cyclosporine A and tacrolimus in experimental liver fibrosis. J Hepatol. 2011 Aug;55(2):388-98. doi: 10.1016/j.jhep.2010.10.044. Epub 2010 Dec 17. PMID 21168455